CLINICAL TRIAL: NCT00254189
Title: A Single Center, Open-Label Study to Evaluate the Effects on Ovulation of Levonorgestrel 90mg and Ethinyl Estradiol 20mg in a Daily, Continuous, Oral Regimen.
Brief Title: Study Evaluating Effects of Levonorgestrel and Ethinyl Estradiol on Ovulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0858A2-208
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2006-05-19 (Estimated); Status verified 2006-05

CONDITIONS: Ovulation
Keywords: Ovulation; Oral Contraceptive
MeSH Terms: interventions — Levonorgestrel; Ethinyl Estradiol

INTERVENTIONS:
Drug: Levonorgestrel
Drug: Ethinyl Estradiol

SUMMARY:
To determine the ability of a monophasic oral contraceptives ("OC") regimen of Levonorgestrel ("LNG") 90 mg and Ethinyl Estradiol ("EE") 20 mg to inhibit ovulation during 84 days of continuous therapy.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of legal age of consent who are willing to use a combination OC.
* Subjects must be under the age of 36 at the time of enrollment (visit 3).
* Subjects must have had regular (24 to 32 day) menstrual cycles for the 3-month period preceding entry into the pretreatment observation cycle, excluding postabortal and nonnursing postpartum subjects. Postabortal and nonnursing postpartum subjects must have completed at least 1 regular (24 to 32 day) spontaneous menstrual cycle before entry into the pretreatment observation cycle. The pretreatment observation cycle for all subjects will begin on day 1 of the subsequent spontaneous menses.

Other inclusions apply.

Exclusion Criteria:

A history or the presence of any of the following will prevent enrollment:

* Thrombophlebitis, thrombosis, or thromboembolic disorders.
* Deep vein thrombosis.
* Pulmonary embolism.

Other exclusions apply.

Ages: 0 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2002-12; Study Completion 2004-10

PRIMARY OUTCOMES:
To determine the ability of a monophasic oral contraceptive (OC) regimen of Levonorgestrel 90 mg and Ethinyl Estradiol 20 mg to inhibit ovulation during 84 days of continuous therapy.

SECONDARY OUTCOMES:
To assess the safety profile. To assess the ovarian activity, as measured by the Hoogland and Skouby 6-point grading system, during 84 days of continuous therapy. To evaluate the time to return of ovulation after cessation of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Archer DF, Kovalevsky G, Ballagh SA, Grubb GS. Ovarian activity and safety of a novel levonorgestrel/ethinyl estradiol continuous oral contraceptive regimen. Contraception. 2009 Sep;80(3):245-53. doi: 10.1016/j.contraception.2009.03.006. Epub 2009 May 2. PMID 19698816